CLINICAL TRIAL: NCT06620393
Title: Effects of Dexmedetomidine on Agitation in Critically Ill TBI Patients (DEX-TBI)
Brief Title: Effects of Dexmedetomidine on Agitation in Critically Ill TBI Patients
Acronym: DEX-TBI
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Canadian Critical Care Trials Group (Other)
Responsible Party: Principal Investigator, David Williamson, Full Clinical Professor, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-32-2024-2732
Record Dates: First submitted 2024-08-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Traumatic Brain Injury; Agitation,Psychomotor
MeSH Terms: conditions — Brain Injuries, Traumatic; Psychomotor Agitation | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): DEX (4 mcg/100 ml supplied by Juno Pharmaceuticals) will be initiated at a starting dose of 0.6 mcg/kg/hour and increased by 0.2 mcg/kg/hour every 30 minutes up to final dose of 1.4 mcg/kg/hour.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Matching placebo (NS 0.9% 100ml)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — DEX 4 mcg/100 ml at a starting dose of 0.6 mcg/kg/hour and increased by 0.2 mcg/kg/hour every 30 minutes up to final dose of 1.4 mcg/kg/hour.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Placebo — NaCl 0.9% 100ml
  Arms: Placebo

SUMMARY:
Agitation is a frequent complication following traumatic braing injury in patients admitted to the intensive care unit. This agitation frequently results in the liberal use of rescue drugs such as antipsychotics, sedatives and opiates, which in turn may delay rehabilitation, liberation from mechanical ventilation and emergence from posttraumatic amnesia. Dexmedetomidine may be a better agent given it's light sedative properties. The main objective is to assess the feasibility of conducting a multicenter randomized controlled trial of dexmedetomidine following TBI in the ICU.

DETAILED DESCRIPTION:
Following a traumatic brain injury, agitation is reported in 53-57% of patients in the intensive care unit. As it is associated with accidental removal of catheters, tubes and dressings as well as self-extubation, agitation poses a threat to patient safety. In addition, agitation can be accompanied by aggressive behaviors that pose a threat to clinician safety. This agitation frequently results in the liberal use of rescue drugs such as antipsychotics, sedatives and opiates, which in turn may delay rehabilitation, liberation from mechanical ventilation and emergence from posttraumatic amnesia. Dexmedetomidine is a highly selective alpha-2 adrenergic receptor agonist used for sedation and also has co-analgesic and withdrawal syndrome alleviating properties. Unlike other sedatives, patients remain easily roused when under dexmedetomidine, facilitating contact and removal from mechanical ventilation. In addition, dexmedetomidine does not induce respiratory depression in critically ill patients. The addition of dexmedetomidine may have the potential to reduce the incidence agitation while reducing the use of agitation rescue drugs such as antipsychotics, the use of physical restraints, as well as the time to cessation of mechanical ventilation and consequently, reduce the time to emergence for post-traumatic amnesia. Duration of posttraumatic amnesia is an important outcome as it is a predictor of cognitive and functional outcomes as well as community integration, psychosocial functioning and employment. The main objective is to assess the feasibility of conducting a multicenter randomized controlled trial of dexmedetomidine following TBI in the ICU. To evaluate the feasibility of conducting a large trial and to refine study procedures, a multicenter randomized double-blind placebo-controlled pilot study comparing dexmedetomidine to placebo will be conducted. The feasibility outcomes will include protocol adherence, trial recruitment and time-in-motion evaluation for study procedures. Clinical outcomes will include agitation, exposure to antipsychotics, time to emergence from post-traumatic amnesia, physical restraint use, ventilator days, and time to ICU and hospital discharge as well as ICU and hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) admitted to ICU with a critically ill moderate or severe TBI patients. Severity of TBI will be determined with the first Glasgow Coma Score (GCS). TBI patients with polytrauma and patients undergoing neurosurgical interventions will be eligible.
2. Undergoing mechanically ventilation (of any duration) at the time of assessment.
3. Anticipated ICU stay of 48 hours or more.

Exclusion Criteria:

1. Patients at very high risk of short-term mortality (e.g., GCS of 3 without sedation, or unreactive pupils, or declared brain-dead when assessed for eligibility and patients in whom there is a lack of commitment to ongoing life support
2. Patients unable to communicate in English or French (interfering with posttraumatic amnesia assessments)
3. Patients with cognitive impairment as per family evaluation
4. Pregnant or breastfeeding
5. Patients currently receiving DEX or clonidine
6. Allergy, bradycardia or hypotension precluding use of dexmedetomidine as per treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Protocol adherence | Through study completion, an average of 2 years
  Proportion of hours the drug was administered

SECONDARY OUTCOMES:
Trial recruitment | Through study completion, an average of 2 years
  Recruitment rate and randomization/activation process (consent rate, proportion of recruited patients who receive the study drug)
Blinding maintenance | Through study completion, an average of 2 years
  Proportion of intensivists and nurses predicting study group assignment at the end of the study intervention and proportion of patients receiving propofol
Proportion of data collection completed | Through study completion, an average of 2 years
  Data collection completeness for agitation-related events, posttraumatic amnesia and cognitive recovery

OTHER OUTCOMES:
ICU-days free of agitation or coma within 14 days following randomization | During ICU stay up to 14 days
  Number of ICU-days without agitation or coma within 14 days following randomization
Agitation-related event during the ICU stay | Through study completion, an average of 2 years
  Accidental device removal, self-extubation following randomization in the ICU
Proportion of patients and the number of days exposed to antipsychotics, benzodiazepines and physical restraints | Through study completion, an average of 2 years
  Exposure to antipsychotics, benzodiazepines and physical restraints after randomization during ICU stay
Time to mechanical ventilation liberation (extubation), time to ICU and hospital discharge | Through study completion, an average of 2 years
  Time to mechanical ventilation liberation (extubation), time to ICU and hospital discharge
Time to emergence from posttraumatic amnesia | Through study completion, an average of 2 years
  Time from randomisation to emergence from posttraumatic amnesia
Cognitive recovery | Through study completion, an average of 2 years
  Brief cognitive assessment in traumatology (EXACT) score (0-100 points); higher scores reflect better function

IPD SHARING:
Plan to Share IPD: No